CLINICAL TRIAL: NCT03390179
Title: Hyperglycemic Response to Steroid Administration After Noncardiac Surgery in Patients With and Without Diabetes
Brief Title: Hyperglycemic Response and Steroid Administration After Surgery (DexGlySurgery)
Acronym: DexGlySurg
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Principal Investigator, Philippe Cuvillon, PhD, Centre Hospitalier Universitaire de Nīmes
Other Study IDs: CHUNimes
Record Dates: First submitted 2017-12-28; First posted 2018-01-04 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Diabetes; Healthy
Keywords: diabetes; anesthesia; surgery; glucose
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- diabetes: Patient with non insulin diabetes
  Interventions: Drug: Steroid Drug
- control: Patient without diabete
  Interventions: Drug: Steroid Drug

INTERVENTIONS:
Drug: Steroid Drug — mesure of the glucose concentration

SUMMARY:
The hyperglycemic response to surgery and the added effect of low-dose steroids (dexamethasone 4 to 8mg), and whether these differ in diabetics and nondiabetics remain unclear. Therefore, we prospectively evaluate the intraoperative and postoperative serum glucose concentrations in diabetics and nondiabetics that received intravenous steroid administration. This multicentre study include > 250 patients.Primary endpoiunt was glucose concentration at H6 after surgery. Secondary endpoints were glucose concentration at H12 and at H24 and effect of anesthesia (regional anesthesia)

ELIGIBILITY:
Inclusion Criteria:

* elective surgery under anesthesia

Exclusion Criteria:

* < 50 kg
* emergency
* insulin therapy
* cardiac surgery
* refusal
* hyperglycemia> 2g/L

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Diabetes (non insulin) or healthy patient scheduled for surgery under anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2017-09-04 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
glucose concentration | 6-8 hour

SECONDARY OUTCOMES:
glucose concentration | 12 hour
glucose concentraion | 24 hour

CONTACTS AND LOCATIONS:
Locations (1):
- Cuvillon, Nîmes, Gard, France

IPD SHARING:
Plan to Share IPD: No